CLINICAL TRIAL: NCT07255612
Title: A Single-arm, Phase II Study for Bone Marrow Protection, Safety, and Efficacy of Trilaciclib Combined With Eribulin in Locally Advanced or Metastatic Triple-negative Breast Cancer After at Least Two Prior Chemotherapy Regimens
Brief Title: Bone Marrow Protection, Safety, Efficacy of Trilaciclib and Eribulin in Locally Advanced or Metastatic TNBC(Triple-negative Breast Cancer)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xu fei, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PROTECTION
Record Dates: First submitted 2024-08-18; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trilaciclib; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trilaciclib Plus Eribulin (Experimental): Trilaciclib: 240mg/m², intravenous infusion for 30 minutes, and completed within 4 hours before chemotherapy administration on day 1 and day 8, day 21 was 1 cycle; Eribulin: 1.4mg/m², intravenous infusion at day 1 and day 8, with 1 cycle at day 21; Note: Trilaciclib combined with Eribulin was treated for cycles 1-2, and continued use of trilaciclib combined with eribulin was a clinical decision from cycle 3 onwards.The infusion interval between treacilil and subsequent injections should not exceed 4 hours.
  Hematopoietic growth factor, blood transfusion, or platelet transfusion are not allowed during the week prior to the blood test during the subject screening period, and no prophylaxis of any cytogenic subclass drugs (including granulocyte colony stimulating factor, granulocyte giant cell colony co-stimulating factor, and erythropoietin) is allowed during the first cycle.However, it can be used therapeutically and should be used in strict accordance with relevant guidelines.
  Interventions: Drug: Trilaciclib; Drug: Eribulin

INTERVENTIONS:
Drug: Trilaciclib — Each participant receives Trilaciclib(240mg/m², intravenous infusion for 30 minutes, and completed within 4 hours before chemotherapy administration on day 1 and day 8, day 21 was 1 cycle)
Drug: Eribulin — Each participant receives Eribulin(1.4mg/m², intravenous infusion at day 1 and day 8, with 1 cycle at day 21)

SUMMARY:
Triple negative breast cancer (TNBC) has attracted much attention due to its young age of onset, high aggressiveness, lack of clear therapeutic targets and poor clinical prognosis.Eribulin is a novel non-taxane anti-microtubule inhibitor with unique microtubule and non-microtubule anti-tumor mechanism.Myelosuppression is the cause of many cancer chemotherapy-related adverse events, such as infections, sepsis, bleeding, and fatigue, resulting in delayed hospital stays or the need for treatment with hematopoietic growth factors, blood transfusions, and more.In addition, myelosuppression usually leads to a lower dose or longer interval of chemotherapy, which reduces the intensity of chemotherapy and affects the benefit of chemotherapy for patients.Trilaciclib is a highly potent, selective and reversible CDK4/6 inhibitor that protects bone marrow by protecting hematopoietic stem cells and progenitor cells (HSPCs) during systemic chemotherapy.

DETAILED DESCRIPTION:
Four randomized, double-blind clinical trials of treacilil in patients with small cell lung cancer (SCLC) confirmed that Trilaciclib administration in combination with chemotherapy prevented or mitigated chemotherapy-induced myelosuppression.Among them, the G1T28-05 study showed that the administration of Trilaciclib before first-line chemotherapy (carboplatin combined with etoposide) could reduce the duration of severe neutropenia in the first cycle from 4 days to 0 days, and the incidence of severe neutropenia from 49.1% to 1.9%.As the world's first drug designed to reduce chemotherapy-induced myelosuppression by protecting HSPCs, Trilaciclib has demonstrated a significant ability to prevent chemotherapy-mediated multicellular lineage myelosuppression in patients with ES-SCLC.In February 2021, the U.S. Food and Drug Administration (FDA) approved Trilaciclib (COSELA™) to reduce the incidence of chemotherapy-induced myelodepression in adult patients with extensive stage small cell lung cancer prior to receiving a platinum-containing/etoposide regimen or topotecan regimen.

Based on the evidence that Trilaciclib has been approved by the FDA to reduce the incidence of chemotherapy-induced myelopathic depression in adult patients with extensive stage small cell lung cancer prior to receipt of a platinum-containing/etoposide regimen or topotecan regimen, there is encouraging patient outcome improvement observed in study G1T28-04.This Phase II clinical trial was designed to confirm the bone marrow protection and efficacy and safety of Trilaciclib in patients with locally advanced/metastatic TNBC who had previously received at least two chemotherapy regimes prior to treatment with Eribulin.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old , no limitation of gender;
2. locally advanced or metastatic triple-negative breast cancer;
3. have received at least two prior chemotherapy regimens(The recurrence of the last adjuvant chemotherapy is counted one line within 12 months after surgery);
4. At least one measurable lesion according to RECIST version 1.1;
5. The laboratory tests meet the following criteria:

   Hemoglobin: ≥ 100 g / L (female), 110g / L (male) Neutrophil count : ≥2×10^9/L Platelet count: ≥100×10^9/L Creatinine：≤15mg / L or creatinine clearance (CrCl) ≥60 mL/min (Cockcroft-Gault formula); Total bilirubin：≤1.5× upper limit of normal (ULN) Alutamate aminotransferase (ALT) and glutamate aminotransferase (AST)≤ 3 ×ULN or 5 ×ULN (for patients with liver metastases) Albumin: ≥ 30 g / L;
6. Eastern Cooperative Oncology Group (ECOG) score [0-1] points;
7. The expected survival period is ≥3 months;
8. During the screening period, all female with potential fertility must have negative serum pregnancy tests and reliable contraception after signing the informed consent form until 3 months after the last dose;
9. Comprehend and voluntarily sign the informed consent form;

Exclusion Criteria:

1. Diagnosed other malignant disease besides breast cancerwithin 5 years before the first dose (excluding radical skin basal cell carcinoma, skin squamous epithelial carcinoma, and / or radical resection);
2. Main organ function not good enough;
3. Bone marrow invasion;
4. Require combined chemotherapy other than Eribulin;
5. Stroke or cardiovascular and cerebrovascular events within 6 months before enrollment;
6. QTcF > 480 msec ( screening period) and QTcF> 500 msec for patients with ventricular pacemaker implantation;
7. Previous hematopoietic stem cell or bone marrow transplantation;
8. Previous G-CSF treatment in the last 2 weeks;
9. Allergic to the study drug or the ingredients;
10. Any other situation where the researcher considers the patient not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2026-11-04 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of grade 3 neutropenia during cycle 1-2 of chemotherapy treatment | 6 months
  evaluated by CIM related index(Chemotherapy-Induced Myelosuppression) , CTCAE5.0(Common Terminology Criteria for Adverse Events)

SECONDARY OUTCOMES:
Anti-tumor efficacy | 6 months
  Conduct tumor imaging assessments. Baseline imaging examinations should be conducted within 21 days prior to the first dose of study drug, and tumor imaging assessments should be conducted every 6 weeks (±7 days) starting from the first administration of the study drug.
  The results of the efficacy evaluations are categorized into complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), and unevaluable (NE).
  Then calculate the indicators to evaluate the anti-tumor efficacy.
  Indicators includes: Objective response rate (ORR),Disease Control Rate( DCR),Duration of response (DOR), Progression free survival (PFS),Overall survival (OS)
Adverse events, abnormal laboratory tests, etal | 6 months
  Adverse events, abnormal laboratory tests, etal; to evaluate safety and tolerability.
Bone marrow protection | 6 months
  Incidence of grade 3 or 4 thrombocytopenia during cycles 1-2; rate of grade 3 or 4 anemia during cycles 1-2; rate of febrile neutropenia; using rate of granulocyte colony-stimulating factor (G-CSF); rate of platelet transfusion; incidence of red cell infusion (week 5 and beyond); using rate of erythropoietin (ESA); using rate of iron; using rate of recombinant human interleukin-11 and / or thrombopoietin (TPO);
Disease burden(cost) | 6 months
  Treatment-related costs of chemotherapy-induced myelosuppression during cycles 1-2 (registration, bed, care, examination / testing and other costs);
Disease burden(in-stay time) | 6 months
  in-stay of myelosuppression caused by chemotherapy
Disease burden(quality of life) | 6 months
  quality of life during chemotherapy (subject EQ-5D-5L, FACT-L and FACT-An scale score)
Compliance with the chemotherapy regimen | 6 months
  Dose of eribulin; The incidence and dose reduction of eribulin chemotherapy during cycles 1-2 of chemotherapy(if there exists dose reduction) ;incidence and duration of delayed changes in chemotherapy(if there exists delayed changes in chemotherapy); and relative dose intensity of eribulin

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No